CLINICAL TRIAL: NCT02209636
Title: Phosphate Lowering to Treat Vascular Dysfunction in Chronic Kidney Disease
Brief Title: Phosphate Lowering in CKD Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNB-006-13F; CX001030 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2014-07-21; First posted 2014-08-06 (Estimated); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-06

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease
Keywords: hyperphosphatemia; vascular dysfunction; chronic kidney disease; cardiovascular disease; endothelial dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Hyperphosphatemia | interventions — lanthanum carbonate; Ascorbic Acid; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lanthanum carbonate (Experimental): Eligible subjects who are randomly assigned to the experimental arm will receive lanthanum carbonate (1500-4500 mg/day in divided doses) titrated to serum phosphorus levels.
  Interventions: Drug: Lanthanum carbonate; Drug: Ascorbic Acid; Drug: Nitroglycerin; Procedure: Flow-mediated dilation measurement; Procedure: Aortic pulse-wave velocity; Procedure: Endothelial cell collection
- placebo (Placebo Comparator): Eligible subjects who are randomly assigned to the placebo arm will receive placebo tablets (identical to the active lanthanum carbonate tablets) to be taken 3 times daily and titrated to serum phosphorus levels.
  Interventions: Drug: placebo; Drug: Ascorbic Acid; Drug: Nitroglycerin; Procedure: Flow-mediated dilation measurement; Procedure: Aortic pulse-wave velocity; Procedure: Endothelial cell collection

INTERVENTIONS:
Drug: Lanthanum carbonate — Non-calcium containing phosphorus binder
  Other Names: Fosrenol
  Arms: Lanthanum carbonate
Drug: placebo — Table identical to lanthanum carbonate but with no active ingredient
  Arms: placebo
Drug: Ascorbic Acid — Intravenous administration during measurement of flow mediated dilation.
  Other Names: Vitamin C
Drug: Nitroglycerin — Drug that is administered under the tongue that relaxes blood vessels. To be administered during measurement of flow mediated dilation.
Procedure: Flow-mediated dilation measurement — Measurement of the blood flow in the brachial artery, an artery in the upper arm, using ultrasound.
Procedure: Aortic pulse-wave velocity — Measurement of the stiffness of the arteries using a transcutaneous tonometer, a small device placed over the skin over the carotid, brachial, radial and femoral arteries.
Procedure: Endothelial cell collection — Collection of endothelial cells from vein in arm. A flexible wire is inserted through an IV into a forearm vein to collect endothelial cells for further study. This is performed at the baseline visit and and the final study visit.

SUMMARY:
The proposed research is a randomized-controlled trial to determine the effectiveness of reducing serum phosphorus using a phosphate binder, lanthanum carbonate, for improving the function of arteries in adults with moderate to severe chronic kidney disease (CKD). [COMIRB 13-0328] Additionally, it will determine phosphorus balance among adults with CKD and whether there is a difference in phosphorus balance after three months of treatment with lanthanum carbonate. [COMIRB 15-0384]

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major health concern both in the general and Veteran populations. Indeed, the prevalence of CKD in a large Veteran population is 20%. Cardiovascular disease (CVD) is significantly increased in CKD and is an important cause of morbidity and mortality. As much as 80% of all CVD is associated with vascular dysfunction, particularly impaired endothelium-dependent dilation (EDD), measured by brachial artery flow-mediate dilation (FMD), and stiffening of the large elastic arteries, measured by aortic pulse-wave velocity (aPWV). Not surprisingly, patients with CKD demonstrate these dysfunctional vascular phenotypes. Even in early stages of CKD, there is an increase in oxidative stress resulting in structural and functional vascular changes, which, in turn, contributes to vascular dysfunction (impaired EDD and large elastic artery stiffening). In CKD, phosphorus remains within the normal range (2.5-4.5 mg/dL) until late in the disease. However, elevated serum phosphorus, even within the normal range, is associated with impaired EDD and with indirect measures of arterial stiffness. Whether lowering serum phosphorus in patients with CKD will improve EDD and arterial stiffness is unknown. This study is a randomized-controlled trial of lanthanum carbonate, a non-calcium based phosphate binder, to treat vascular dysfunction. The efficacy of phosphate binding with lanthanum carbonate for treating vascular endothelial dysfunction and large elastic artery stiffness in patients with stage IIIb and IV CKD (estimated glomerular filtration rate 15-45 mL/min/1.73m2) with baseline serum phosphorus of 2.8-5.5 mg/dL will be assessed. The study will also determine if lowering serum phosphorus with lanthanum carbonate also reduces circulating and endothelial cell markers of oxidative stress. This study could shift clinical practice guidelines by establishing a novel therapy for reducing CVD risk in CKD patients not requiring chronic hemodialysis. [COMIRB 13-0328]

Little is known about phosphorus balance in CKD. It is assumed that CKD patients remain in neutral phosphorus balance despite decreases in kidney function. Serum phosphorus remains in the normal range until late in CKD thus making it difficult to recognize perturbations in phosphorus balance. Indeed, among CKD patients treated with the non-calcium containing phosphate binder, sevelamer, serum phosphorus did not change after six weeks of treatment but urinary phosphate excretion, parathyroid hormone, and fibroblast growth factor-23 changed significantly, suggesting a shift in phosphorus homeostasis. However, two other studies found that patients with CKD III-IV treated with calcium-containing phosphate binders remained in neutral phosphorus balance. There are no studies evaluating the effects of non-calcium based phosphate binders on phosphorus balance among patients with CKD nor other studies examining the effect of changing phosphorus balance on vascular function.

An extension of the above-described 12-week prospective randomized, placebo-controlled double-blind trial (COMIRB 13-0328) will be conducted in a subset of subjects. A total of 24 subjects from COMIRB 13-0328 will be recruited to participate in the Phosphorus Balance sub-investigation (12 subjects treated with lanthanum carbonate and 12 subjects treated with placebo). [15-0384] They will consume a diet with a fixed phosphorus content (1000 +/- 50 mg) for seven days. They will then be admitted to the inpatient Center for Translational Clinical Research at the University of Colorado Denver for 48 hours to accurately collect urine and stool samples. The goal of the Phosphorus Balance sub-investigation (COMIRB 15-0384) is to determine whether lowering serum phosphorus, accomplished during the parent phosphorus lowering randomized-controlled trial (COMIRB 13-0328), affects phosphorus balance compared to those subjects treated with placebo. A key secondary goal is to determine if differences in phosphorus balance affect vascular function as measured by FMD. [15-0384]

To ensure adequate enrollment in the Phosphorus Balance Study (COMIRB 15-0384), an amendment was approved to recruit patients with stage IIIb and IV CKD with normal or modestly elevated serum phosphorus (2.8-5.5 mg/dL) who are not currently participating in the parent Phosphorus Lowering RCT (COMIRB 13-0328). Similar to the Phosphorus Lowering RCT, these patients will follow a low phosphorus diet and will be randomized to lanthanum carbonate or placebo for 12 weeks (run-in period) prior to beginning the current Phosphorus Balance protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-79, women must be post-menopausal
* CKD stage IIIb or IV (estimated glomerular filtration rate by MDRD 15-45 mL/min/1.73m2), stable for 3 months
* Serum phosphorus 2.8-5.5 mg/dL, stable for 3 months
* Not using phosphate binders
* Albumin > 3.0 g/dL
* Free from alcohol dependence or abuse
* Ability to provide informed consent
* BMI < 40 kg/m2
* Not taking medications that interact with agents administered during experimental sessions (e.g., sildenafil interacts with nitroglycerin)
* For COMIRB 15-0384, completion of the prospective, randomized, placebo-controlled double-blind trial, Phosphorus Lowering to Treat Vascular Dysfunction in Chronic Kidney Disease (COMIRB 13-0328) or completion of 12-week run-in phase

Exclusion Criteria:

* Life expectancy <1 year
* Uncontrolled hypertension
* History of severe liver disease
* History of congestive heart failure (EF < 35%)
* History of hospitalizations within the last 3 months
* History of ileus or bowel obstruction
* Active infection or antibiotic therapy
* Expected kidney transplant in the next 6 months
* Active vitamin D analogue use (i.e. calcitriol, paricalcitol, doxercalciferol)
* Vasculitis requiring immunosuppressive therapy within the last year
* Current tobacco abuse

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna J Jovanovich, MD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jovanovich A, Struemph T, You Z, Wang W, Farmer-Bailey H, Bispham N, Levi M, Schwartz GG, Nowak KL, Chonchol M. Effect of Lanthanum Carbonate on Serum Phosphate, Oxidative Stress, and Vascular Dysfunction in CKD: A Mechanistic Randomized Controlled Trial. Kidney360. 2024 Jul 1;5(7):959-966. doi: 10.34067/KID.0000000000000465. Epub 2024 May 23. PMID 38781013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N = 66 completed screening and signed consent so were considered enrolled; however, N = 5 did not receive allocated intervention because N = 3 withdrew consent, N = 1 had uncontrolled hypertension after screening, and N =1 had phosphorus levels that were too low to receive study drug after screening.
Period: Main/Parent Study
Arm/Group | Lanthanum Carbonate | Placebo
Started | 32 | 29
Completed | 27 | 27
Not Completed | 5 | 2
Period: Balance Sub-study
Arm/Group | Lanthanum Carbonate | Placebo
Started | 7 | 8
Completed | 6 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanthanum Carbonate | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 65 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 27 | 25 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 26 | 26 | 52
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-mediated Dilation
Description: Measurement of how well the brachial artery dilates in response to shear stress. It is a measure of endothelial function. It is reported as "percent change", which represents the change in dilation of the artery before and after occlusion.
  Brachial artery flow-mediated dilation will be measured at baseline and at 12 weeks (end-of-study) in the treatment and placebo groups to determine if there is a change brachial artery flow mediated dilation from baseline to 12 weeks and if this change is significantly different between the treatment and placebo groups.
Time Frame: baseline and 12 weeks
Population: Participants were analyzed if they had baseline and end-of-study FMD measurements and the measurements were of sufficient quality to be analyzed.
Measure: Mean (Standard Deviation); unit: percent change FMD
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 25 | 27
percent change FMD
  baseline | 3.13 (2.87) | 3.74 (2.86)
  week 12 | 2.73 (2.48) | 3.09 (2.49)

2. Primary Outcome: Aortic Pulse-wave Velocity
Description: The speed that blood travels from the carotid artery to the femoral artery, expressed as cm/s (centimeters/second). It is a measure of arterial stiffness.
  Aortic pulse-wave velocity will be measured at baseline and at 12 weeks (end-of-study) in the treatment and placebo groups to determine if there is a change aortic pulse wave velocity from baseline to 12 weeks and if this change is significantly different between the treatment and placebo groups.
Time Frame: baseline and 12 weeks
Population: Participants were included if they had baseline and end of study aPWV measurements and aPWV measurements were of sufficient quality to be analyzed.
Measure: Mean (Standard Deviation); unit: change in aPWV, cm/s
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 25 | 25
change in aPWV, cm/s
  baseline | 1214 (394) | 993 (289)
  week 12 | 1216 (321) | 977 (254)

3. Primary Outcome: Phosphorus Balance Sub-study (COMIRB 15-0384)
Description: Balance is defined as oral intake minus urine output minus stool output.
Time Frame: 9 days from the start of the sub-study, approximately 13 weeks and 2 days from the start of the Main/Parent Study
Population: Subjects who participated in the Phosphorus Balance sub-study and had sufficient stool volume for analysis.
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 6 | 8
mg/d | -131 (163) | 320 (141)

4. Secondary Outcome: Oxidative Stress-associated Suppression of EDD
Description: The influence of oxidative stress on FMD will be determined by infusing a supraphysiologic dose of ascorbic acid or isovolemic saline. The difference in FMD, expressed as percentage change in FMD, which represents the change in dilation of the artery before and after occlusion, during ascorbic acid vs. saline infusion will be taken as a measure of the modulation of EDD/stiffness by oxidative stress.
Time Frame: baseline and 12 weeks
Population: Participants were included if they had baseline and end of study FMD measurements, FMD measurements were of sufficient quality to be analyzed, and were able to receive ascorbic acid infusion.
Measure: Mean (Standard Deviation); unit: percent change in FMD
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 22 | 24
percent change in FMD
  baseline FMD: number analyzed (Participants) | 21 | 24
  baseline FMD | 2.91 (2.81) | 3.54 (2.86)
  baseline FMD after ascorbic acid: number analyzed (Participants) | 21 | 24
  baseline FMD after ascorbic acid | 3.24 (3.48) | 3.44 (2.70)
  week 12 FMD: number analyzed (Participants) | 21 | 24
  week 12 FMD | 2.48 (2.54) | 2.95 (2.10)
  week 12 FMD w/ ascorbic acid: number analyzed (Participants) | 21 | 24
  week 12 FMD w/ ascorbic acid | 3.44 (3.19) | 3.69 (3.03)

5. Secondary Outcome: Vascular Endothelial Cell Protein Expression
Description: Measures of different protein markers on endothelial cells. Will help understand the underlying pathophysiology of vascular dysfunction in chronic kidney disease. Vascular endothelial cell protein expression will be measured at baseline and at 12 weeks (end-of-study) in the treatment and placebo groups to determine if there is a change vascular endothelial cell protein expression from baseline to 12 weeks and if this change is significantly different between the treatment and placebo groups. The expression of endothelial cells collected from patients will be compared to the expression in HUVEC (human umbilical vein endothelial cell) controls and this ratio will be reported as the outcomes measure.
Time Frame: baseline and 12 weeks
Population: Participants with sufficient number of collected endothelial cells for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 17 | 14
ratio
  baseline | 1.54 (0.31) | 1.41 (0.25)
  week 12 | 1.44 (0.26) | 1.40 (0.15)

6. Secondary Outcome: Interleukin-6 to Measure Systemic Inflammation
Description: This is a blood test. Interleukin-6 and C-reactive protein will be measured at baseline and at 12 weeks (end-of-study) in the treatment and placebo groups to determine if there is a change in interleukin-6 and C-reactive protein from baseline to 12 weeks and if this change is significantly different between the treatment and placebo groups.
Time Frame: baseline and 12 weeks
Population: Participants were included if they had baseline and end of study blood collected.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 27 | 27
pg/ml
  Interleukin-6, baseline | 1.58 [1.06 to 2.36] | 1.28 [0.93 to 2.20]
  Interleukin-6, week 12 | 1.61 [1.12 to 2.56] | 1.34 [0.88 to 2.68]

7. Secondary Outcome: Oxidized Low-density Lipoprotein (Ox-LDL) to Measure Systemic Oxidized Stress
Description: This is a blood test art. Oxidized low-density lipoprotein (ox-LDL) will be measured at baseline and at 12 weeks (end-of-study) in the treatment and placebo groups to determine if there is a change in ox-LDL from baseline to 12 weeks and if this change is significantly different between the treatment and placebo groups.
Time Frame: baseline and 12 weeks
Population: Participants were included if they had blood collected at baseline and end of study.
Measure: Median (Inter-Quartile Range); unit: mU/ml
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 27 | 27
mU/ml
  baseline | 61837 [49168 to 81461] | 62927 [49634 to 82774]
  week 12 | 59725 [48650 to 86949] | 68057 [52199 to 78069]

8. Secondary Outcome: C-reactive Protein to Measure Systemic Inflammation
Description: This is a blood test. C-reactive protein will be measured at baseline and at 12 weeks (end-of-study) in the treatment and placebo groups to determine if there is a change in C-reactive protein from baseline to 12 weeks and if this change is significantly different between the treatment and placebo groups.
Time Frame: baseline and 12 weeks
Population: Participants were included if they had baseline and end of study blood collected.
Measure: Median (Inter-Quartile Range); unit: mg/ml
Arm/Group | Lanthanum Carbonate | Placebo
Number analyzed (Participants) | 27 | 27
mg/ml
  C-reactive protein, baseline | 2.92 [1.36 to 6.61] | 2.72 [1.06 to 5.95]
  C-reactive protein, week 12 | 3.06 [1.02 to 5.93] | 2.24 [1.18 to 3.95]

ADVERSE EVENTS:
Time Frame: 12 weeks (i.e., study duration for each participant in the Main/Parent Study); 9 days (i.e., study duration of Phosphorus Balance Sub-study)
Groups:
- Lanthanum Carbonate- Phosphorus Balance Sub-study: Continued randomized intervention from Parent/Main Study on and received a fixed phosphorus diet for 9 days after the completion of the Parent/Main Study.
- Placebo- Phosphorus Balance Sub-study: Continued randomized intervention from Parent/Main Study on and received a fixed phosphorus diet for 9 days after the completion og the Parent/Main Study.
Arm/Group | Lanthanum Carbonate | Placebo | Lanthanum Carbonate- Phosphorus Balance Sub-study | Placebo- Phosphorus Balance Sub-study
All-Cause Mortality (participants affected / at risk) | 1/32 | 0/29 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/32 | 1/29 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 12/32 | 4/29 | 0/7 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate (N=32) | Placebo (N=29) | Lanthanum Carbonate- Phosphorus Balance Sub-study (N=7) | Placebo- Phosphorus Balance Sub-study (N=8)
Hospitalization (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for hepatic encephalopathy
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Hospitalization for pneumonia.
Hospitalization (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for cerebral vascular accident (CVA) (i.e., stroke).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate (N=32) | Placebo (N=29) | Lanthanum Carbonate- Phosphorus Balance Sub-study (N=7) | Placebo- Phosphorus Balance Sub-study (N=8)
Non-serious adverse events (Gastrointestinal disorders) | 12 (19) | 4 (4) | 0 (0) | 0 (0) — Constipation, diarrhea, nausea, vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT02209636/Prot_SAP_000.pdf